CLINICAL TRIAL: NCT00421720
Title: A Randomized, Open-label, Multicenter, Parallel-group Study to Compare the Efficacy, Safety and Resource Utilization of a Remifentanil/Propofol Analgesia/Sedation Regimen Versus a Sufentanil/Propofol Analgesia/Sedation Regimen in Mechanically Ventilated Intensive Care Patients Requiring Analgesia and Sedation for up to 7 Days
Brief Title: A Study Comparing Two Analgesia/Sedation Regimens, Remifentanil/Propofol Versus Sufentanil/Propofol In Mechanically Ventilated Intensive Care Patients Requiring Analgesia And Sedation.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USA107212; EudraCT: 2006-001276-20
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Analgesia; Sedation
Keywords: remifentanil; sufentanil; propofol; analgesia; sedation; mechanically ventilated; intensive care; pharmacoeconomic; weaning; delirium; randomized; Germany
MeSH Terms: conditions — Agnosia; Delirium | interventions — Sufentanil; Remifentanil

INTERVENTIONS:
Drug: Sufentanil
Drug: Remifentanil

SUMMARY:
This prospective, randomized, multicenter, open-label study will compare two analgesia-based regimens for sedation (remifentanil/propofol vs. sufentanil/propofol) in medium to long-term ventilated intensive care patients in terms of efficacy, safety and resource utilization.

The special characteristics of intensive care patients (organ insufficiencies etc.) regularly cause an accumulation of the analgesics, sedatives and adjuvants used. Clinically, this complicates the calculation of weaning and extubation times, often making mechanical ventilation necessary for longer periods than desired and also extending the stay of patients in the intensive care unit. Reducing weaning times and the duration of intensive care treatment by optimizing analgesia/sedation could furthermore lead to a reduction in typical complications such as ventilator-associated pneumonia or delirium.

The demands on an ideal analgesic are analgesic efficacy without severe cardiopulmonary depression and rapid onset of effect and in particular a short dura-tion of effect and absence of accumulation or development of active metabolites. Remifentanil is an ultra-short acting µ-agonist which is, due to its molecular structure, metabolized organ-independently by unspecific blood and tissue esterases with the substance being degraded within only a few minutes and the resulting metabolites being virtually ineffective at the µ-receptor. Sufentanil, on the other hand, is mainly metabolized by the cytochrome P-450-3A4 enzyme in the liver and small intestine.

To date, only one study with a small sample size is available on the comparison of the effectiveness and safety of remifentanil and sufentanil when used for long-term analgesia/sedation.

ELIGIBILITY:
INCLUSION CRITERIA

* Written informed consent was obtained from the patient
* The patient is under intensive medical care, intubated and ventilated
* The expected duration of ventilation and analgesia/sedation is > 24 hours and </= 7 days
* Propofol is planned to be used as sedative

EXCLUSION CRITERIA

* Contraindication against administration of remifentanil, sufentanil, or propofol
* Concomitant medications:
* The patient is receiving epidural analgesia or a peripheral regional anesthetic therapy.
* The patient is requiring muscle relaxants to facilitate mechanical ventilation
* The patient participated in clinical drug trials within the previous 30 days or participated in this clinical trial before or is currently participating in any other clinical trial
* The patient has a known hypersensitivity to the drugs under investigation or to propofol (and other components of the preparation to be used), soy and peanut
* For female patients: the patient is pregnant or breastfeeding
* The patient is classified as ASA V or moribund
* The patient must be expected to show an impaired cerebral or neurologic capacity due to illness, trauma or other interventions, which will interfere with the collection of the analgesia/sedation scores and the waking behavior as for example, without being limited to:
* Hypoxic brain damage
* Cerebrocranial trauma grades II, III, and IV
* Subarachnoid hemorrhage, brain-stem hemorrhage, ischemic-hemorrhagic cerebral hemorrhages
* Amyotrophic lateral sclerosis, myasthenia gravis
* Stupor or coma
* The patient requires chronic ventilation
* The patient is receiving chronic (> 3 months) therapy with high-potency opioids/WHO level 3
* The patient is alcohol or drug dependent (legal or illegal drugs in particular, but not exclusively with dependency on sedatives or benzodiazepines), defined as:
* Typically an urgent desire to take the substance, problems in controlling consumption, and persistent use of the substance despite adverse consequences. The use of the substance has priority over other activities and responsibilities. Developing increased tolerance and occasionally physical withdrawal symptom.
* The patient suffers from a manifest organ failure
* The patient suffers from severe heart failure, NYHA Class IV (symptoms at rest)
* The patient has a history of or actually suffers from ventricular tachycardia, ventricular flutter or ventricular fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164
Dates: Start 2007-01

PRIMARY OUTCOMES:
Comparison of ventilation and weaning times: - Time from initiation of analgesia/sedation using the investigational substance and extubation ("ventilation time") - Time from the start of weaning to extubation ("weaning time")

SECONDARY OUTCOMES:
ICU length of stay; accuracy of analgesia/sedation; drug consumption of analgesics/sedatives; clinical course; incidence of pneumonia/delirium; infection markers; bowel movement; ventilation parameters; vital signs; resource utilization; safety

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, PhD, Study Director — GlaxoSmithKline
Locations (10):
- Germany (10):
  - GSK Clinical Trials Call Center, Bonn
  - GSK Clinical Trials Call Center, Dresden
  - GSK Clinical Trials Call Center, Heidelberg
  - GSK Clinical Trials Call Center, Homburg/Saar
  - GSK Clinical Trials Call Center, Kiel
  - GSK Clinical Trials Call Center, Ludwigshafen
  - GSK Clinical Trials Call Center, Rostock
  - GSK Clinical Trials Call Center, Saarbrücken
  - GSK Clinical Trials Call Center, Schwerin
  - GSK Clinical Trials Call Center, Tübingen